CLINICAL TRIAL: NCT06820047
Title: Impact of Sleeve Gastrectomy Versus Intensive Lifestyle Modifications With Obesity Management Medications on BMI Trajectory and Target Attainment: a Prospective Matched Cohort Study
Brief Title: Sleeve Gastrectomy vs. Lifestyle & Medications: Impact on BMI Trajectory and Target Attainment in a Matched Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Lidia Castagneto Gissey, Prof, University of Roma La Sapienza
Other Study IDs: ID3361963
Record Dates: First submitted 2025-01-27; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Obesity-related Medical Conditions
Keywords: obesity; sleeve gastrectomy; semaglutide; glp-1 receptor agonist; intensive lifestyle modifications
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Surgical Group: Patients undergoing laparoscopic sleeve gastrectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- Medical Group: Patients undergoing intensive lifestyle modifications + semaglutide 2.4 mg once weekly
  Interventions: Other: Obesity pharmacotherapy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Patients underwent SG, involving longitudinal resection of approximately 75% of the stomach along its greater curvature, with excision of the fundus and part of the body and antrum, preserving a portion of the latter and the pylorus itself. This results in a vertical tube-shaped gastric tube "sleeve". After surgery, patients followed a free diet. Patients were evaluated at baseline and at 1, 3, 6, 9, and 12 months after starting the intervention.
  Groups: Surgical Group
Other: Obesity pharmacotherapy — Patients underwent 1 month of a very low calorie diet (VLCD) with 813 kcal/day, followed by a low calorie diet (LCD) for 11 months together with intensive physical exercise (30 min/day of brisk walking plus at least 3 h/week of aerobic exercise) with 2.4 mg/week of semaglutide (Ozempic®), given once weekly as subcutaneous injections. Patients were evaluated at baseline and at 1, 3, 6, 9 and 12 months after starting the interventions.
  Other Names: Intensive Lifestyle Modifications; Semaglutide 2.4 mg
  Groups: Medical Group

SUMMARY:
Obesity is a widespread and preventable condition affecting over a billion people globally, with rates expected to rise significantly by 2030. It increases the risk of chronic illnesses such as diabetes, cardiovascular disease, certain cancers, mental health issues, and premature death. While bariatric surgery, such as sleeve gastrectomy (SG), is the most effective long-term weight-loss solution, many individuals are ineligible or unwilling to undergo surgery. Semaglutide, a medication that suppresses appetite and aids in weight loss when paired with diet and exercise, offers a promising alternative. This study compared the effectiveness of SG and an intensive weight-loss program combining diet, exercise, and semaglutide. Conducted over a year with 190 participants split into two groups matched by BMI, the SG group underwent surgery, while the other group followed a calorie-restricted diet, intensive exercise, and weekly semaglutide injections. Changes in BMI, weight, and comorbidities such as diabetes and high blood pressure were evaluated, aiming to determine which approach was more effective in managing obesity.

DETAILED DESCRIPTION:
Obesity is a complex and largely preventable disease affecting over a third of the global population. As of 2022, more than 1 billion individuals worldwide were living with obesity, and projections indicate that by 2030, 38% of the adult population will be overweight, with an additional 20% affected by obesity. This condition significantly increases the risk of chronic diseases, including type 2 diabetes (T2D), cardiovascular disease (CVD), certain cancers, and mental health disorders such as depression, as well as premature mortality.

Given the rising prevalence of obesity, effective intervention strategies are critical. Bariatric and metabolic surgery remains the most effective approach for sustained weight loss, with procedures recommended for individuals with a body mass index (BMI) ≥35 kg/m², regardless of comorbidities. Metabolic surgery has demonstrated superior outcomes in reducing blood glucose levels and achieving higher remission rates of T2D compared to lifestyle and pharmacological interventions. However, surgical interventions are typically reserved for individuals who have failed prior dietary and exercise-based interventions, have adequate motivation, and do not suffer from severe psychiatric conditions.

For individuals who are ineligible for or unwilling to undergo bariatric surgery, alternative treatment options are necessary. One such option is semaglutide, a glucagon-like peptide-1 (GLP-1) receptor agonist, which mimics endogenous GLP-1 to suppress appetite, reduce glucagon release, and promote satiety. Studies have shown that GLP-1 receptor agonists contribute to significant weight loss and metabolic improvements.

This study aims to compare the efficacy of intensive lifestyle modifications combined with obesity management medications (ILM/OMMs) versus sleeve gastrectomy (SG) in terms of BMI trajectory and metabolic outcomes over a 1-year period. The primary endpoint is the change in BMI at 1 year, while secondary endpoints include changes in weight, plasma glucose levels, lipid profiles, and obesity-related comorbidities such as hypertension, CVD, dyslipidemia, and T2D.

Methods Study Design This study is a 1-year, prospective, multicenter, matched cohort study comparing ILM/OMMs with SG. Patients were recruited from the weight-loss clinics of Sapienza University Hospital and Catholic University Hospital in Rome, Italy. Eligible patients were allocated to either ILM/OMMs or SG. Ninety-five patients per arm were matched in a 1:1 ratio, based on sex, age, BMI, and diabetes duration.

The study was conducted between May 2022 and July 2024, following the STROBE (STrengthening the Reporting of OBservational studies in Epidemiology) reporting guidelines for cohort studies. Ethical approval was obtained from both institutions, and the study was conducted in accordance with the Declaration of Helsinki and Good Clinical Practice guidelines. Written informed consent was obtained from all participants, with additional consent required for patients undergoing bariatric surgery.

Participants

Inclusion criteria:

Age 19-69 years Stable body weight for the past 6 months BMI ≥35 kg/m² with at least one obesity-related comorbidity (T2D, hypertension, sleep apnea, metabolic-associated fatty liver disease, osteoarthritis, dyslipidemia, gastrointestinal disorders, or heart disease) or BMI ≥40 kg/m²

Exclusion criteria:

Previous bariatric surgery History of pancreatitis Severe psychiatric disorders Personal or familial history of endocrine cancers

Interventions Medical Arm (ILM/OMMs Group) Participants underwent a 1-month very low-calorie diet (VLCD) of 813 kcal/day, followed by an 11-month low-calorie diet (LCD), combined with structured physical activity (30 minutes/day of brisk walking and at least 3 hours/week of aerobic exercise). Additionally, they received 2.4 mg/week of semaglutide (Ozempic®) administered as a subcutaneous injection. Clinical evaluations were conducted at baseline and at 1, 3, 6, 9, and 12 months.

Surgical Arm (SG Group) Patients underwent SG, a procedure involving the longitudinal resection of approximately 75% of the stomach along its greater curvature, including the excision of the fundus, part of the body, and antrum while preserving the pylorus. Following surgery, patients were allowed a free diet. Clinical evaluations were performed at baseline and at 1, 3, 6, 9, and 12 months.

Outcome Measures The primary endpoint was the change in BMI at 1 year and the time required to achieve a 25% reduction in BMI. Secondary endpoints included changes in weight, plasma glucose levels, lipid profiles, and obesity-related comorbidities such as hypertension, CVD, dyslipidemia, and T2D at 1 year from baseline.

Body weight and height were measured using calibrated scales with participants wearing light clothing. The percentage of total body weight loss was calculated using the formula:

Sample Size Calculation To determine equivalence between the surgical and ILM/OMMs groups, the study was powered to detect a true mean difference of 3% in weight loss (25% in ILM/OMMs vs. 28% in SG) with an equivalence margin of 5%. Assuming a standard deviation of 3.4%, a sample size of 76 patients per group (alpha = 0.05, power = 90%) was required. Considering a 20% attrition rate, the final sample size was set at 190 patients (95 per group).

Statistical Analysis To assess treatment equivalence in percentage weight loss, a t-test was performed. Changes in clinical outcomes were analyzed using t-tests or Mann-Whitney U tests for continuous variables and chi-squared or Fisher's exact tests for categorical variables. Logistic regression models were used to compare response curves for weight loss and comorbidity resolution, adjusting for covariates. Continuous data were expressed as mean ± standard deviation (SD), while categorical variables were presented as counts and percentages. All statistical analyses were performed using SPSS Statistics v.27.0

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 69 years with stable body weight in the past 6 months;
* BMI ≥35 kg/m2 and at least one or more obesity-related co-morbidities (T2D, hypertension, sleep apnea and other respiratory disorders, metabolic-associated fatty liver disease, osteoarthritis, lipid abnormalities, gastrointestinal disorders, or heart disease)
* BMI≥40 kg/m2 with or without related comorbidities

Exclusion Criteria:

* Previous bariatric surgery;
* History of pancreatitis;
* Severe psychiatric disorders;
* Personal or familiar history of endocrine cancers.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the weight-loss clinic of Sapienza University Hospital and Catholic University Hospital in Rome, Italy, and eligible for bariatric surgery were allocated to intensive lifestyle modifications with obesity management medications or metabolic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Weight modifications | 12 months
  Change in body mass index (expressed as weight in kilograms divided by height in meters squared, kg/m^2) at 1 year and time to reach 25% total weight loss (%TWL) (weight will be reported in kilograms)

SECONDARY OUTCOMES:
Glycemic control changes | 12 months
  - Plasma glucose (in mg/dL)
Lipid profile changes | 12 months
  Lipid profile (in mg/dL) changes
Comorbidity resolution rate | 12 months
  Hypertension remission rate (in percentage)
Comorbidity resolution rate | 12 months
  Type 2 diabetes remission rate (in percentage)
Comorbidity resolution rate | 12 months
  Dyslipidemia remission rate (in percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Castagneto Gissey, MD, PhD, Study Director — University of Roma La Sapienza
Locations (2):
- Italy (2):
  - IRCCS Catholic University of Rome, Rome, Italy
  - Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request at lidia.castagnetogissey@uniroma1.it
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 1 month and ending 10 years after the publication of results
Access Criteria: IPD will be shared with qualified researchers conducting scientifically valid analyses relevant to obesity management and metabolic interventions. Access to the data will require submission of a research proposal outlining the planned analyses and statistical methods. Proposals must be reviewed and approved by an independent data access committee. A formal data-sharing agreement must be signed before access is granted. Requests can be submitted via the institutional research office at Sapienza University Hospital via email (lidia.castagnetogissey@uniroma1.it). Data access decisions will be based on scientific merit, ethical considerations, and compliance with data protection regulations.